CLINICAL TRIAL: NCT07011732
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled, Parallel Group Study to Evaluate the Safety and Efficacy of KarXT + KarX-EC for the Treatment of Agitation Associated With Alzheimer's Disease
Brief Title: A Phase 3 Study to Evaluate the Safety and Efficacy of KarXT + KarX-EC for the Treatment of Agitation Associated With Alzheimer's Disease (ADAGIO-1)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CN012-0023; 2025-520613-31 (Other: EU CTR); U1111-1316-5745 (Other: WHO)
Record Dates: First submitted 2025-06-02; First posted 2025-06-10 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — xanomeline; trospium chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- KarXT + KarX-EC (Experimental)
  Interventions: Drug: Xanomeline/Trospium Chloride Capsule; Drug: Xanomeline Enteric Capsule
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Xanomeline/Trospium Chloride Capsule — Specified dose on specified days
  Other Names: KarXT; BMS-986510
  Arms: KarXT + KarX-EC
Drug: Xanomeline Enteric Capsule — Specified dose on specified days
  Other Names: KarX-EC; BMS-986519
  Arms: KarXT + KarX-EC
Drug: Placebo — Specified dose on specified days
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of KarXT + KarX-EC in adult participants with agitation related to Alzheimer's Disease.

ELIGIBILITY:
Inclusion Criteria

- A diagnosis of Alzheimer's disease (AD) in accordance with the 2024 Alzheimer's Association criteria with one of the following confirmations of AD pathology: i) Historical evidence of AD diagnosis with amyloid positron emission tomography (PET), Aβ42/40 ratio in CSF, pTau181/Aβ42 ratio in CSF or pTau217/Aβ42 ratio in plasma using an Health Authority (HA)-authorized diagnostic assay.

ii) If no historical evidence available: A. A plasma biomarker will be assessed for eligibility if allowed per regulatory requirements. The test cutoff(s) will be based on diagnostic use approval.

B. If a plasma biomarker assay cannot be used or if the assay result is inconclusive, conduct one the following:

* Amyloid PET.
* Aβ42/40 ratio or pTau181/Aβ42 ratio in CSF using an HA-authorized diagnostic assay.

  * Mini-Mental State Examination (MMSE) score of 5 to 22, inclusive, at Screening (Visit 1).
  * Have one identified caregiver who should have sufficient contact (approximately 10 hours a week or more) and is willing to:

    i) Attend all visits and report on participant's status. ii) Oversee participant compliance with medication and study procedures. iii) Participate in the study assessments and provide informed consent to participate in the study.
  * History of agitation that meets the International Psychogeriatric Association (IPA) consensus definition for agitation in cognitive disorders with onset at least two weeks prior to Screening (Visit 1).
  * AD participants are required to have NPI/NPI-NH Agitation/Aggression score ≥ 4 at Screening (Visit 1) and Baseline (Visit 2).
  * CGI-S ≥ 4, as related to agitation, at Screening (Visit 1) and Baseline (Visit 2).
  * At least 1 of the following 3 criteria must be established from the CMAI-IPA at Screening (Visit 1) and Baseline (Visit 2; CMAI-IPA Physical/Verbal Aggression Positivity):

    i) 1 or more aggressive behaviors occurring at least several times per week. ii) 2 or more aggressive behaviors occurring at least once or twice per week. iii) 3 or more aggressive behaviors occurring less than once per week.

Exclusion Criteria

- Medical Conditions: i) Agitation symptoms that are primarily attributable to a condition other than the AD causing the dementia.

ii) History of bipolar disorder, schizophrenia, or schizoaffective disorder. iii) History of (or at high risk for) urinary retention, gastric retention, or narrow-angle glaucoma as evaluated by the Investigator.

iv) Risk of suicidal behavior during the study as determined by the Investigator's clinical assessment and/or C-SSR.

- Prior/Concomitant Therapy: i) Recent history of receiving monoamine oxidase inhibitors, anticonvulsants (eg, lamotrigine, divalproex), mood stabilizers (eg, lithium), tricyclic antidepressants (eg, imipramine, desipramine), or any other psychoactive medications except for as needed anxiolytics (eg, lorazepam).

A. Selective serotonin reuptake inhibitors and serotonin norepinephrine reuptake inhibitors taken at a stable dose for at least 8 weeks prior to Screening (Visit 1) may be permitted.

B. Mirtazapine or trazodone may be used as a hypnotic if started at least 8 weeks prior to Screening (Visit 1).

- Other protocol-defined Inclusion/Exclusion criteria apply.

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 352 (Estimated)
Dates: Start 2025-07-10 (Actual); Primary Completion 2028-11-24 (Estimated); Study Completion 2028-12-08 (Estimated)

PRIMARY OUTCOMES:
Change from baseline on the Cohen-Mansfield Agitation Inventory-International Psychogeriatric Association (CMAI-IPA) total score at Week 14 | At Week 14

SECONDARY OUTCOMES:
Change from baseline on the Clinical Global Impressions-Severity (CGI-S) at Week 14 | At Week 14
Change from baseline on the CMAI-IPA Domains at Week 14 | At Week 14
Change from baseline on the CMAI Total Score at Week 14 | At Week 14
Number of participants with Occurrence of Response at Week 14 | At Week 14
  As determined by CMAI-IPA changes of at least 30%, 40%, and 50% from baseline
Change from baseline on the Neuropsychiatric Inventory/Neuropsychiatric Inventory -Nursing Home (NPI/NPI-NH) Total Score at Week 14 | At Week 14
Number of participants with Adverse Events (AEs) | Up to Week 18
Number of participants with Treatment Emergent AEs (TEAEs) | Up to Week 18
Number of participants with Serious AEs (SAEs) | Up to Week 18
Number of participants with AEs leading to study drug withdrawal | Up to Week 18
Number of deaths | Up to Week 18
Number of participants with AEs of Special Interest (AESIs) | Up to Week 18
Barnes Akathisia Rating Scale (BARS) | Up to Week 18
Abnormal Involuntary Movement Scale (AIMS) | Up to Week 18
Body Weight | Up to Week 18
Body Mass Index (BMI) | Up to Week 18
Number of participants with vital sign abnormalities | Up to Week 18
Number of participants with clinical laboratory abnormalities | Up to Week 18
Number of participants with electrocardiogram (ECG) abnormalities | Up to Week 18
Number of participants with suicidal ideation as assessed by the Columbia-Suicide Severity Rating Scale (C-SSRS) | Up to Week 18
Severity of benign prostatic hyperplasia in male participants as assessed by International Prostate Symptom Score (IPSS) | Up to Week 18

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (155):
- United States (42):
  - Imaging Endpoints, Scottsdale, Arizona
  - Advanced Research Center (ARC) - Anaheim, Anaheim, California
  - Kaizen Brain Center, La Jolla, California
  - The Neurology Group, Pomona, California
  - Torrance Clinical Research, Torrance, California
  - Sunwise Clinical Research, Walnut Creek, California
  - Local Institution - 1630, Colorado Springs, Colorado
  - Local Institution - 1622, Maitland, Florida
  - Local Institution - 1631, Maitland, Florida
  - Local Institution - 1602, Miami, Florida
  - Local Institution - 1618, Miami, Florida
  - Hope Research Network - Miami, Miami, Florida
  - Nuovida Research Center, Miami, Florida
  - Local Institution - 1608, Ocala, Florida
  - Combined Research Orlando (CRO), Orlando, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Local Institution - 1661, Savannah, Georgia
  - Local Institution - 1655, Marrero, Louisiana
  - CBH Health, Gaithersburg, Maryland
  - Local Institution - 1663, Foxborough, Massachusetts
  - Boston Center for Memory, Newton, Massachusetts
  - Mayflower Clinical Research, South Dartmouth, Massachusetts
  - Local Institution - 1660, Springfield, Massachusetts
  - Local Institution - 1665, Bloomfield Hills, Michigan
  - Oakland Medical Research, Troy, Michigan
  - Redbird Research, Las Vegas, Nevada
  - Patient First MD, Middletown, New Jersey
  - Local Institution - 1664, Princeton, New Jersey
  - Local Institution - 1610, Inwood, New York
  - Mid Hudson Medical Research, New Windsor, New York
  - Local Institution - 1645, Woodmere, New York
  - Local Institution - 1658, Woodmere, New York
  - Local Institution - 1601, Monroe, North Carolina
  - Local Institution - 1659, Centerville, Ohio
  - Central States Research, Tulsa, Oklahoma
  - Local Institution - 1652, Columbia, South Carolina
  - Local Institution - 1653, Columbia, South Carolina
  - Advanced Neurology Epilepsy and Sleep Center, El Paso, Texas
  - Wasatch Clinical Research, LLC, Salt Lake City, Utah
  - Local Institution - 1646, Bennington, Vermont
  - Local Institution - 1644, Seattle, Washington
  - Kingfisher Cooperative, Spokane, Washington
- Argentina (7):
  - Local Institution - 1001, La Plata, Buenos Aires
  - Local Institution - 1002, Mar del Plata, Buenos Aires
  - Local Institution - 1006, Rosario, Santa Fe Province
  - Local Institution - 1003, Buenos Aires
  - Local Institution - 1004, Córdoba
  - Instituto Privado Kremer, Córdoba
  - Local Institution - 1000, Córdoba
- Brazil (9):
  - Local Institution - 1051, Brasília, Federal District
  - Local Institution - 1052, Curitiba, Paraná
  - Local Institution - 1053, Curitiba, Paraná
  - Local Institution - 1058, Porto Alegre, Rio Grande do Sul
  - Local Institution - 1054, Porto Alegre, Rio Grande do Sul
  - Local Institution - 1057, Campinas, São Paulo
  - Local Institution - 1056, São Paulo, São Paulo
  - Local Institution - 1050, Rio de Janeiro
  - CPQuali Pesquisa Clínica, São Paulo
- Bulgaria (4):
  - Local Institution - 1100, Sofia, Sofia-Grad
  - Local Institution - 1101, Pleven
  - Outpatient Clinic for Individual Practice for Specialized Medical Care in Psychiatry - Dr. Madlena Dimitrova Borisova, Razgrad
  - Medical Center Mladost, Varna
- Canada (7):
  - Local Institution - 1153, Hamilton, Ontario
  - Local Institution - 1155, London, Ontario
  - Local Institution - 1755, London, Ontario
  - Sunnybrook Research Institute, Toronto, Ontario
  - Local Institution - 1154, Toronto, Ontario
  - Ontario Shores Centre For Mental Health Sciences, Whitby, Ontario
  - Local Institution - 1150, Montreal, Quebec
- China (17):
  - Local Institution - 1805, Beijing, Beijing Municipality
  - Local Institution - 1810, Beijing, Beijing Municipality
  - Local Institution - 1815, Haidian District, Beijing Municipality
  - Local Institution - 1813, Chongqing, Chongqing Municipality
  - Local Institution - 1809, Guangzhou, Guangdong
  - Local Institution - 1802, Guangzhou, Guangdong
  - Local Institution - 1818, Shenzhen, Guangdong
  - Local Institution - 1803, Changsha, Hunan
  - Local Institution - 1801, Nanjing, Jiangsu
  - Local Institution - 1800, Shanghai, Shanghai Municipality
  - Local Institution - 1816, Xian, Shanxi
  - Local Institution - 1819, Chengdu, Sichuan
  - Local Institution - 1814, Tianjin, Tianjin Municipality
  - Local Institution - 1804, Hangzhou, Zhejiang
  - Local Institution - 1817, Hangzhou
  - Local Institution - 1812, Kunming
  - Local Institution - 1808, Tianjin
- Croatia (5):
  - Local Institution - 1550, Zagreb, City of Zagreb
  - Local Institution - 1553, Zagreb, City of Zagreb
  - Local Institution - 1554, Rijeka
  - Local Institution - 1551, Split
  - Local Institution - 1552, Varaždin
- Greece (8):
  - Local Institution - 1200, Pátrai, Achaḯa
  - Local Institution - 1205, Athens, Attica
  - Local Institution - 1202, Athens, Attica
  - Aiginiteio University Hospital, Athens, Attikí
  - University General Hospital "ATTIKON" - General Hospital of West Attica "H AGIA VARVARA", Chaïdári, Attikí
  - Local Institution - 1207, Athens
  - Local Institution - 1201, Ioannina
  - Local Institution - 1204, Thessaloniki
- India (7):
  - Local Institution - 1251, Hyderabad, Andhra Pradesh
  - Local Institution - 1255, Ahmedabad, Gujarat
  - Local Institution - 1252, Hyderabad, Telangana
  - Local Institution - 1254, Varanasi, Uttar Pradesh
  - Local Institution - 1250, Kolkata, West Bengal
  - Local Institution - 1256, Delhi
  - Local Institution - 1253, New Delhi
- Japan (9):
  - Local Institution - 1301, Hadano, Kanagawa
  - Teikyo University Mizonokuchi Hospital, Kawasaki, Kanagawa
  - Local Institution - 1304, Sakai, Osaka
  - National Hospital Organization Hizen Psychiatric Center, Kanzaki-Gun Yoshinogari-Cho, Saga-ken
  - Rainbow and Sea Hospital, Karatsu-shi, Saga-ken
  - Local Institution - 1305, Bunkyo-ku, Tokyo
  - Kuramitsu Hospital, Fukuoka
  - Local Institution - 1306, Okayama
  - Local Institution - 1308, Shimotsuke-shi, Tochigi
- Mexico (9):
  - Local Institution - 1355, Saltillo, Coahuila
  - Boca Clinical Trials Mexico S.C., Guadajalara, Jalisco
  - Local Institution - 1364, Monterrey, Nuevo León
  - Local Institution - 1350, Monterrey, Nuevo León
  - Local Institution - 1361, Mexico City
  - Local Institution - 1363, Mexico City
  - Local Institution - 1360, Mexico City
  - Local Institution - 1362, San Luis Potosí City
  - Clinical Research Institute S.C., Tlalnepantla
- Portugal (5):
  - Local Institution - 1401, Coimbra
  - Centro Hospitalar do Alto Ave, Guimarães
  - Local Institution - 1404, Lisbon
  - Unidade Local de Saúde de Matosinhos SA, Senhora da Hora
  - Campus Neurologico Senior, Torres Vedras
- Romania (10):
  - Local Institution - 1450, Bucharest, București
  - Local Institution - 1453, Bucharest, București
  - Local Institution - 1454, Bucharest, București
  - Prof. Dr. Alexandru Obregia Psychiatry Hospital, Bucharest, București
  - Local Institution - 1451, Bucharest
  - Local Institution - 1459, Bucharest
  - Local Institution - 1461, Constanța
  - Local Institution - 1457, Iași
  - Local Institution - 1460, Sanpetru /Brasov
  - Local Institution - 1462, Sibiu
- Spain (11):
  - Oroitu Centro de Atencion Especializada, Getxo, Bizkaia
  - Hospital General Universitario de Elche, Elche (alicante)
  - Complejo Hospitalario Ruber Juan Bravo, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Clinico Universitario Virgen de La Victoria, Málaga
  - Local Institution - 1507, Pamplona
  - Hospital Universitario de Salamanca - Complejo Asistencial Universitario de Salamanca, Salamanca
  - Hospital Victoria Eugenia de Sevilla, Seville
  - Hospital Mutua Terrassa, Terrassa
  - Hospital Universitario De Rio Hortega, Valladolid
  - Hospital Viamed Montecanal, Zaragoza
- Taiwan (5):
  - Local Institution - 1753, Kaohsiung Niao Sung Dist, Kaohsiung
  - National Cheng Kung University Hospital, Tainan, Taiana
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Medical Foundation-Linkou Branch, Taoyuan District

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT07011732.html